CLINICAL TRIAL: NCT02431624
Title: A Two Period, Randomised, Open-label, Crossover Study to Assess the Adhesion of Buprenorphine Transdermal Delivery System 40 µg/h Patch and 20 µg/h Patch, in Healthy Volunteers
Brief Title: An Assessment of Buprenorphine Transdermal Delivery System (BTDS) Patch Adhesion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BUP1508; 2014-003421-18 (EudraCT Number)
Record Dates: First submitted 2015-02-25; First posted 2015-05-01 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Pain
Keywords: Healthy Volunteer
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test treatment (Experimental): BTDS 40 milligram
  Interventions: Drug: BTDS
- Reference treatment (Active Comparator): BTDS 20 milligram
  Interventions: Drug: BTDS

INTERVENTIONS:
Drug: BTDS

SUMMARY:
The purpose of this study is to assess the adhesion of BTDS patch 40 µg/h.

DETAILED DESCRIPTION:
The objective is to show non-inferiority in adhesion of BTDS patch 40 µg/h compared to BTDS patch 20 µg/h. Safety and tolerability of both patches will also be assessed.

ELIGIBILITY:
1. Provide written informed consent.
2. Healthy male or female subjects aged 18 to 55 inclusive.
3. Female subjects of child bearing potential must be willing to use two highly effective methods of contraception throughout the study, one of which must include a barrier method.
4. Female subjects who are postmenopausal (defined as spontaneous amenorrhoea for at least 1 year) or permanently sterilised (e.g. tubal occlusion, hysterectomy, bilateral salpingectomy). These subjects are not required to use any contraception.
5. Male subjects who are willing to use contraception with their partners throughout the study and for 30 days after completion of the study and agree to inform the Investigator if their partner becomes pregnant during this time.
6. Body weight ranging from 55 to 100 kg and a BMI ≥ 18.5 and ≤ 30.0.
7. Healthy and free of significant abnormal findings as determined by medical history, physical examination, vital signs, laboratory tests and ECG.
8. The subject's primary care physician has confirmed within the last 12 months of first dosing that there is nothing in the subject's medical history that would preclude their enrolment into a clinical study.

Exclusion Criteria

Subjects to be excluded from the study are those who meet any of the following criteria:

1. Female subjects who are pregnant or lactating.
2. Any history of drug or alcohol abuse.
3. Any history of conditions that might interfere with drug absorption, distribution, metabolism or excretion.
4. Use of opioid or opioid antagonist-containing medication in the past 30 days.
5. Any history of frequent nausea or vomiting regardless of aetiology.
6. Any history of seizures or symptomatic head trauma.
7. Participation in a clinical drug study during the 90 days preceding the initial dose in this study, or participation in any other clinical drug study during this study.
8. Any significant illness during the 4 weeks preceding entry into this study.
9. A history of additional risk factors for Torsades de Pointes (e.g. heart failure, hypokalaemia, personal or family history of long QT syndrome, syncope, or family history of sudden death).
10. Abnormal cardiac conditions including any of the following:

    * QTcF interval greater than 450 msec at screening or at check-in before first dosing.
    * Increase in QTcF of more than 60 msec above pre-dose values of each study period or QTcF > 500 msec at any time during the study.
11. Use of medication within 5 times the half-life or minimum 14 days for prescription medication or 7 days for over-the-counter preparations (including vitamins, herbal and/or mineral supplements), whichever is longer, before the first dose of study treatment and during the study (with the exception of the continued use of Hormone Replacement Therapy (HRT) and contraceptives).
12. Refusal to abstain from caffeine or xanthine containing beverages and grapefruit juice within 48 hours before IMP administration until after the last study measure has been performed in each study period.
13. Weekly alcohol intake exceeding the equivalent of 14 units/week for females and 21 units/week for males.
14. Consumption of alcoholic beverages within 48 hours before IMP administration, and refusal to abstain from alcohol for the duration of the study confinement and for at least 48 hours after the last naltrexone dose in each study period.
15. History of smoking within 45 days of IMP administration and refusal to abstain from smoking during the study.
16. Positive results of urine drug screen, alcohol test and pregnancy test.
17. Known sensitivity to buprenorphine, naltrexone, related compounds or any of the excipients or any contraindications as detailed in the Butrans Summary of Product Characteristics or Nemexin Summary of Product Characteristics.
18. Clinically significant history of allergic reaction to wound dressings or elastoplast.
19. Subjects with any dermatological disorder or tattoos at the proposed sites of patch application, or with a history of eczema/cutaneous atrophy.
20. Subjects who will not allow hair to be removed at the proposed patch application sites which may prevent proper placement of the patch.
21. Refusal to allow their primary care physician to be informed of participation in the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patch Adhesion score | 7 days

SECONDARY OUTCOMES:
Observer Rating Scale of Patch prior to Removal questionnaire | 7 days
  does the patch shift, buckle, curl, fall off, change colour or smell
Skin reaction assessment score | day 8
Adverse Events | Up to 7-10 days post patch removal
Changes in haematology and biochemistry values | Up to 7-10 days after last patch removal
Vital signs | Up to 7-10 days after last patch removal
ECG | Up to 7-10 days after last patch removal

CONTACTS AND LOCATIONS:
Locations (1):
- BioKinetic Europe Ltd, Belfast, United Kingdom